CLINICAL TRIAL: NCT00919802
Title: Intranasal Oxytocin for the Treatment of Pain Associated With Interstitial Cystitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Tim Ness, MD, MD, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UAB0001
Record Dates: First submitted 2009-06-09; First posted 2009-06-12 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial cystitis (IC); Oxytocin; Bladder; Void
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Active Comparator): Oxytocin, 40 IU intranasally, once
  Interventions: Drug: Oxytocin
- Saline as a nasal spray (Placebo Comparator): Saline, 4ml intranasally, once
  Interventions: Other: Saline as a nasal spray

INTERVENTIONS:
Drug: Oxytocin — A single dose of oxytocin 40 IU (20 IU to each nostril) will be dispensed in a random fashion to subjects. A log will be kept so that the subject will receive a single does of saline as an alternate agent on the second day if needed.
  Other Names: Syntocinon
  Arms: Oxytocin
Other: Saline as a nasal spray — A single dose of saline will be dispensed in a random fashion to subjects. A log will be kept so that the subject will receive a single does of oxytocin 40 IU as an alternate agent on the second day if needed.
  Arms: Saline as a nasal spray

SUMMARY:
Anecdotal evidence suggests female patients with painful bladder disorder interstitial cystitis (IC) can experience a significant attenuation of their systems while breastfeeding. Since it has been shown that postpartum lactation is a time associated with decreased levels of stress, and stress has been shown to exacerbate IC-related pain, the investigators have developed an interest in the effects of the hormones involved in postpartum lactation on stress and pain. Based on a series of pre-clinical experiments, the investigators believe the hormone oxytoxin has both analgesic and anxiolytic properties which make it a potentially useful agent for the treatment of stress-exacerbated chronic pain syndrome such as IC. Therefore, the investigators propose a double-blinded, placebo-controlled crossover trial of intranasal oxytocin vs. intranasal saline for bladder pain in a cohort of patients with IC and some degree of continuous, daily pain.

DETAILED DESCRIPTION:
Fifty patients will be enrolled in a double-blinded, placebo-controlled single-dose crossover trial comparing intranasal oxytocin to intranasal saline. At the time of enrollment, patients will complete a series of standardized questionnaires detailing information about their IC-related symptoms at baseline as well as comorbid conditions, coping mechanisms (specifically catastrophizing), and baseline ratings of overall pain, depression, anxiety, and global functioning. Once this information is obtained, the patient will receive a one-time dose of intranasal oxytocin or an equivalent volume of intranasal saline. The patients will be monitored for one hour by a physician investigator for toxicities and efficacy and then contacted for follow-up information at 2, 4, 6, and 24 hours. At each of these time points, the patient will be asked to report a verbal pain report, a verbal anxiety report, the number of voids since last contact with an investigator, and the use of any additional medications for pain control or anxiety. In addition, a global response assessment (GRA) score will be obtained at 6 and 24 hours. The patient will be asked to return within a one week period at which time he/she will receive the alternative intranasal agent. Following the second dose, the patient will be monitored for one hour and contact made at 2, 4, 6, and 24 hours as previously described.

The primary outcome measure will be the GRA score, which will be analyzed using a Chi-square analysis followed by Fischer's exact test. Secondary outcome measures will be analyzed via ANOVA.

If this study indicates that intranasal oxytocin is efficacious for pain control, this could provide for an alternative to current ineffective or invasive treatments for IC-related pain. It is also possible it could eventually be utilized for other forms of chronic pain as well.

ELIGIBILITY:
Inclusion Criteria:

* 19 - 65 years of age
* Must meet the current National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) diagnostic criteria for interstitial cystitis and have some degree of continuous daily pain

Exclusion Criteria:

* Pregnancy
* Under the age of 19
* Older that the age of 65
* Breastfeeding women
* Uncontrolled hypertension
* History of significant cardiac or pulmonary disease (including arrhythmias)
* Known allergy to oxytocin
* Severe psychiatric disease
* Patients who have undergone procedural interventions within the past month related to their interstitial cystitis

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith T Robbins, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified raw data will be made available on request by contacting contact investigator at tness@uabmc.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: June 2010, Primary Completion Date: September 2015 and Study Completion Date: September 2015. Recruitment location: University of Alabama at Birmingham.
Pre-assignment Details: The major goal of this project was to evaluate the efficacy of intranasal oxytocin in relieving bladder pain in a cohort of patients with interstitial cystitis.
Groups:
- Intranasal Oxytocin, Followed by Intranasal Saline: Oxytocin, 40 IU intranasally, once
  Oxytocin: A single dose of oxytocin 40 IU (20 IU to each nostril) will be dispensed in a random fashion to subjects. Patients will be monitored for one hour by a physician investigator for toxicities and efficacy, and then contacted for follow-up information at 2, 4, 6 and 24 hours. The patient will be asked to return within a one-week period at which time the patient will receive the alternative intranasal agent. Following the second dose, the patient will be monitored for one hour and contact made at 2, 4, 6, and 24 hours as previously described.
- Intranasal Saline Followed With Intranasal Oxytocin: Saline, 4ml intranasally, once
  Patients will be randomized to receive saline as a nasal spray: A single dose of saline will be dispensed in a random fashion to subjects.
  Patients will be monitored for one hour by a physician investigator for toxicities and efficacy, and then contacted for follow-up information at 2, 4, 6 and 24 hours. The patient will be asked to return within a one-week period at which time they will receive the alternative intranasal agent, Oxytocin a single dose of oxytocin 40 IU (20 IU to each nostril). Following the second dose, the patient will be monitored for one hour and contact made at 2, 4, 6, and 24 hours as previously described.
Period: First Intervention - (24 Hours)
Arm/Group | Intranasal Oxytocin, Followed by Intranasal Saline | Intranasal Saline Followed With Intranasal Oxytocin
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0
Period: Second Intervention - (24 Hours)
Arm/Group | Intranasal Oxytocin, Followed by Intranasal Saline | Intranasal Saline Followed With Intranasal Oxytocin
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Patients will be randomized to receive a single dose of oxytocin 40 IU (20 IU to each nostril) or saline. Patients will be monitored for one hour by a physician investigator for toxicities and efficacy, and then contacted for follow-up information at 2, 4, 6 and 24 hours. The patient will be asked to return within a one-week period at which time the patient will receive the alternative intranasal agent. Following the second dose, the patient will be monitored for one hour and contact made at 2, 4, 6, and 24 hours as previously described.
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Measured as Global Response Assessment (GRA) Score at 6 and 24 Hours
Description: This is a seven-point symmetric scale previously validated for use in IC studies in which patients are asked relative to baseline (over the last 6 hours for purposes of this study), -3 -are you markedly worse, -2 -moderately worse, -1 -slightly worse, 0-no change, +1-slightly improved, +2-moderately improved, or +3-markedly improved. A +2 or +3 can be defined categorically as a positive treatment response
Time Frame: 6 and 24 hours post drug or placebo administration - the data below reflects 6 hour data
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oxytocin | Saline as a Nasal Spray
Number analyzed (Participants) | 25 | 25
units on a scale | .5 (.2) | -.1 (.2)
Statistical Analysis 1: Comparison: Oxytocin vs Saline as a Nasal Spray; Global Response Assessment (GRA) scores were obtained 6 and 24 hours post oxytocin or saline administration; Test type: Other; p = 0.688, t-test, 2 sided

2. Secondary Outcome: Secondary Outcome Measures Will Include Change From Baseline in Verbal Reports of Anxiety 6 Hours After Drug/Placebo Administration
Description: A verbal anxiety report (VAR; 0-10 with 0 being no anxiety and 10 being the worst possible anxiety); a change from baseline measure was calculated for value measured 6 hours post drug/placebo administration
Time Frame: 6 hours post drug or placebo administration
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oxytocin | Saline as a Nasal Spray
Number analyzed (Participants) | 25 | 25
units on a scale | -1.2 (.4) | -1.0 (.4)
Statistical Analysis 1: Comparison: Oxytocin vs Saline as a Nasal Spray; Test type: Other — paired t-test comparison of change in VAR from baseline 6 hours after drug; a change in VAR score was calculated for each subject for each arm and compared using a paired t-test; p = 0.7252, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for 24 hours after each drug/placebo administration
Description: Patients did not report any adverse events
Arm/Group | Oxytocin | Saline as a Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No